CLINICAL TRIAL: NCT02424188
Title: Trial of Integrated Smoking Cessation, Exercise and Weight Management in Serious Mental Illness: TRIUMPH
Acronym: TRIUMPH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Massachusetts General Hospital (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00072510; R01MH104553 (NIH)
Record Dates: First submitted 2015-04-18; First posted 2015-04-22 (Estimated); Results first posted 2025-06-25 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Mental Illness
Keywords: weight management; physical activity; Tobacco smoking; Serious mental illness
MeSH Terms: conditions — Mental Disorders; Motor Activity; Tobacco Smoking

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TRIUMPH intervention (Experimental): Group and individual smoking cessation and weight management counseling, pharmacotherapy with varenicline or bupropion and nicotine replacement therapy, group exercise, and text messaging support
  Interventions: Other: TRIIUMPH Intervention
- Treatment as Usual (No Intervention): referral to quit line

INTERVENTIONS:
Other: TRIIUMPH Intervention — Group and individual smoking cessation and weight management counseling, pharmacotherapy with varenicline or bupropion and nicotine replacement therapy, group exercise, and text messaging support
  Arms: TRIUMPH intervention

SUMMARY:
This study will determine whether an 18-month practical tobacco smoking cessation program integrating weight management counseling and exercise will be superior to treatment as usual in achieving prolonged smoking abstinence in persons with serious mental illness.

DETAILED DESCRIPTION:
The objective of this study is to perform a randomized clinical trial (TRIUMPH) in persons with serious mental illness to test the hypothesis that intervention participants will have higher rates of smoking abstinence at 18 months than participants in the treatment as usual arm. The intervention includes group and individual smoking cessation and weight management counseling tailored by a participant's readiness to quit, pharmacotherapy with either varenicline or buproprion plus nicotine replacement therapy prescribed in the community clinic, exercise, and text messaging supporting health behavior change.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia, schizoaffective disorder, bipolar disorder, or recurrent major depression meeting criteria for serious mental illness
* Fagerstrom Test for Nicotine Dependence of ≥3 and daily cigarette smoking for at least the past 6 months (on days that cigarettes were available)
* On stable psychotropic medication for mental illness for at least 30 days (i.e., antipsychotic medication for those with schizophrenia spectrum illness, mood stabilizer for those with bipolar disorder)
* Competent and willing to give informed consent
* Completion of baseline data collection
* Willing to participate in smoking cessation intervention that includes combination of evidence-based behavioral (group and individual sessions) and pharmacotherapeutic smoking cessation aids

Exclusion Criteria:

* Serious cardiovascular event (e.g. myocardial infarction, stroke) within the past 6 months
* Serious unstable medical condition that limits life expectancy
* Pregnant, breastfeeding, or planning a pregnancy during study period.
* Alcohol or illicit substance use disorder if not sober/abstinent for ≥ 30 days
* Planning to leave mental health program or move out of geographic area within 18 months Review by treating psychiatrist required for those with inpatient psychiatric hospitalization within six months of enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2016-07-07 (Actual); Primary Completion 2020-03 (Actual); Study Completion 2020-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gail L Daumit, MD, MHS, Principal Investigator — Johns Hopkins University; A. Eden Evins, MD, MPH, Principal Investigator — Massachussetts General Hospital
Locations (1):
- Johns Hopkins, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Daumit GL, Evins AE, Cather C, Dalcin AT, Dickerson FB, Miller ER 3rd, Appel LJ, Jerome GJ, McCann U, Ford DE, Charleston JB, Young DR, Gennusa JV 3rd, Goldsholl S, Cook C, Fink T, Wang NY. Effect of a Tobacco Cessation Intervention Incorporating Weight Management for Adults With Serious Mental Illness: A Randomized Clinical Trial. JAMA Psychiatry. 2023 Sep 1;80(9):895-904. doi: 10.1001/jamapsychiatry.2023.1691. PMID 37378972

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | TRIUMPH Intervention | Treatment as Usual
Started | 97 | 95
Completed | 93 | 90
Not Completed | 4 | 5
Not completed — Death | 2 | 2
Not completed — Lost to Follow-up | 1 | 3
Not completed — Incarceration | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TRIUMPH Intervention | Treatment as Usual | Total
Number analyzed (Participants) | 97 | 95 | 192
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 89 | 86 | 175
  >=65 years | 8 | 9 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 48 (12.1) | 51.3 (11) | 49.6 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 52 | 97
  Male | 52 | 43 | 95
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 3 | 6
  Not Hispanic or Latino | 93 | 92 | 185
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 47 | 46 | 93
  White | 45 | 45 | 90
  More than one race | 4 | 2 | 6
  Unknown or Not Reported | 1 | 1 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 97 | 95 | 192
Primary Psychiatric Diagnosis [Count of Participants; unit: Participants]
  Schizophrenia | 12 | 15 | 27
  Schizoaffective disorder | 30 | 25 | 55
  Bipolar disorder | 29 | 33 | 62
  Major depressive disorder | 26 | 22 | 48
Smoking, Willingness to quit [Count of Participants; unit: Participants]
  Quit in 2 months | 61 | 58 | 119
  Quit in 6 months | 36 | 37 | 73
Fagerstrom Test for Nicotine Dependence [Mean (Standard Deviation); unit: scores on a scale] — Total score range of 0-10 (0=minimum to 10=maximum nicotine dependence), higher score is worse
  scores on a scale | 4.5 (2) | 4.6 (2) | 4.5 (2)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Smoking Abstinence
Description: 7-day point prevalence, biochemically validated
Time Frame: measured at 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | TRIUMPH Intervention | Treatment as Usual
Number analyzed (Participants) | 97 | 95
Participants | 27 | 6
Statistical Analysis 1: Comparison: TRIUMPH Intervention vs Treatment as Usual; Test type: Superiority; Odds Ratio (OR) = 5.9, 95% CI 2-sided [2.3 to 15.4]

2. Secondary Outcome: Smoking Abstinence - 3 Months
Description: Participants with 3 month smoking abstinence
Time Frame: from 15 to 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | TRIUMPH Intervention | Treatment as Usual
Number analyzed (Participants) | 97 | 95
Participants | 14 | 4
Statistical Analysis 1: Comparison: TRIUMPH Intervention vs Treatment as Usual; Test type: Superiority; Odds Ratio (OR) = 3.9, 95% CI 2-sided [1.2 to 12.3]

3. Secondary Outcome: Smoking Abstinence
Description: 7-day point prevalence, biochemically validated
Time Frame: measured at 6 and 12 months
Measure: Count of Participants; unit: Participants
Arm/Group | TRIUMPH Intervention | Treatment as Usual
Number analyzed (Participants) | 97 | 95
Participants
  6 month: abstinent | 13 | 3
  6 month: not abstinent | 84 | 92
  12 month: abstinent | 18 | 2
  12 month: not abstinent | 79 | 93
Statistical Analysis 1: Comparison: TRIUMPH Intervention vs Treatment as Usual; 6 month comparison; Test type: Superiority; Odds Ratio (OR) = 4.8, 95% CI 2-sided [1.3 to 17.5]
Statistical Analysis 2: Comparison: TRIUMPH Intervention vs Treatment as Usual; 12 month; Test type: Superiority; Odds Ratio (OR) = 10.8, 95% CI 2-sided [2.4 to 48.6]

4. Secondary Outcome: 12 Months Continuous Smoking Abstinence
Description: participants who reported smoking abstinence continuously from 6 months 18 months
Time Frame: measured from 6 months to 18 months
Measure: Count of Participants; unit: Participants
Arm/Group | TRIUMPH Intervention | Treatment as Usual
Number analyzed (Participants) | 97 | 95
Participants
  Abstinent | 6 | 0
  Not abstinent | 91 | 95

5. Secondary Outcome: Weight
Description: weight in kilograms
Time Frame: Baseline, 6 and 18 months
Measure: Mean (95% Confidence Interval); unit: kilograms
Arm/Group | TRIUMPH Intervention | Treatment as Usual
Number analyzed (Participants) | 97 | 95
kilograms
  Baseline | 92.1 [87.6 to 96] | 89.8 [85.3 to 94.3]
  6 month | 92.2 [87.6 to 96] | 89.6 [84.9 to 94.4]
  18 month | 92.2 [87.4 to 97] | 88.4 [83.4 to 93.3]
Statistical Analysis 1: Comparison: TRIUMPH Intervention vs Treatment as Usual; 6 months; Test type: Superiority; Mean Difference (Net) = 0.3, 95% CI 2-sided [-1.7 to 2.3]
Statistical Analysis 2: Comparison: TRIUMPH Intervention vs Treatment as Usual; 18 months; Test type: Superiority; Mean Difference (Net) = 1.6, 95% CI 2-sided [-1.5 to 4.7]

6. Secondary Outcome: Body Mass Index
Time Frame: Baseline, 18 months
Measure: Mean (Standard Deviation); unit: kg/m^2
Arm/Group | TRIUMPH Intervention | Treatment as Usual
Number analyzed (Participants) | 97 | 95
kg/m^2
  Baseline | 32.1 (8.2) | 32 (7)
  18 months | 32.3 (8.9) | 31.3 (7.3)
Statistical Analysis 1: Comparison: TRIUMPH Intervention vs Treatment as Usual; Test type: Superiority; Mean Difference (Net) = 0.4, 95% CI 2-sided [-0.6 to 1.5]

7. Secondary Outcome: Six Minute Walk
Time Frame: 18 months
Population: A substantial proportion of the follow-up visits were off-site where the standardized six-minute walk course could not be used.
Measure: Mean (Standard Deviation); unit: feet
Arm/Group | TRIUMPH Intervention | Treatment as Usual
Number analyzed (Participants) | 87 | 82
feet
  Baseline | 1000.7 (403.1) | 943.8 (321.5)
  18 month | 953.6 (208.2) | 942.4 (384.1)

8. Secondary Outcome: Framingham Stroke Risk Profile Score
Description: The score can range from 0-38 with higher scores yielding increased 10-year probability of stroke
Time Frame: 18 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TRIUMPH Intervention | Treatment as Usual
Number analyzed (Participants) | 97 | 95
score on a scale
  Baseline | 9.5 (2.6) | 11.1 (2.9)
  18 months | 9.3 (2.7) | 11.6 (2.7)
Statistical Analysis 1: Comparison: TRIUMPH Intervention vs Treatment as Usual; Test type: Superiority; Mean Difference (Net) = -16.2, 95% CI 2-sided [-30.2 to -2.3]

9. Secondary Outcome: Health Status as Assessed by the Short Form -12 (SF-12) Index
Description: SF-12 Mental Health Index and Physical Composite (scores range from 0-100), the higher the score means a better outcome
Time Frame: 6 and 18 months
Population: No modeled
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TRIUMPH Intervention | Treatment as Usual
Number analyzed (Participants) | 97 | 95
score on a scale
  physical score-baseline | 45.0 (10.6) | 43.2 (10.3)
  physical score-6 month | 45.5 (8.6) | 42.5 (10.5)
  physical score-18 month | 45.8 (9.2) | 43.1 (8.2)
  mental score- baseline | 46.8 (7.6) | 45.5 (9.6)
  mental score- 6 month | 48.3 (9.2) | 46.2 (10.3)
  mental score- 18 month | 48.3 (7.9) | 48.0 (8.6)

10. Secondary Outcome: Psychiatric Symptoms Assessed by the Brief Psychiatric Rating Scale
Description: Brief Psychiatric Rating Scale. Total scores range from a minimum score of 18 to a maximum score of 126. A higher total score indicates a more severe psychiatric symptom rating.
Time Frame: Baseline
Population: Data not collected at follow up due to excessive participant burden and insufficient staff needed to maintain adequate inter-rater reliability at follow-up time points.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TRIUMPH Intervention | Treatment as Usual
Number analyzed (Participants) | 93 | 90
score on a scale | 42.0 (12.5) | 41.0 (10.7)

ADVERSE EVENTS:
Time Frame: Up to 18 months
Arm/Group | TRIUMPH Intervention | Treatment as Usual
All-Cause Mortality (participants affected / at risk) | 2/97 | 2/95
Serious Adverse Events (participants affected / at risk) | 31/97 | 23/95
Other Adverse Events (participants affected / at risk) | 0/97 | 0/95
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TRIUMPH Intervention (N=97) | Treatment as Usual (N=95)
Psychiatric hospitalization (Psychiatric disorders) | 11 (13) | 9 (11)
Medical hospitalization (General disorders) | 20 (23) | 16 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-29): https://cdn.clinicaltrials.gov/large-docs/88/NCT02424188/Prot_SAP_000.pdf